CLINICAL TRIAL: NCT00827177
Title: A Phase 1 Dose Escalation Study of ARQ 197 in Combination With Sorafenib in Adult Patients With Advanced Solid Tumors
Brief Title: Dose Escalation Study of ARQ 197 in Combination With Sorafenib in Adult Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ArQule, Inc., a subsidiary of Merck Sharp & Dohme LLC, a subsidiary of Merck & Co., Inc. (Rahway, NJ USA) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARQ 197-116
Record Dates: First submitted 2009-01-21; First posted 2009-01-22 (Estimated); Last update posted 2014-01-24 (Estimated); Status verified 2014-01

CONDITIONS: Advanced Solid Tumors
Keywords: dose escalation; safety; tolerability; tumor; PK; hepatocellular carcinoma; renal cell carcinoma; melanoma; non-small cell lung cancer; breast cancer
MeSH Terms: conditions — Neoplasms; Carcinoma, Hepatocellular; Carcinoma, Renal Cell; Melanoma; Carcinoma, Non-Small-Cell Lung; Breast Neoplasms | interventions — Therapeutics; ARQ 197; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ARQ 197 in combination with sorafenib (Experimental)
  Interventions: Drug: Treatment with ARQ 197 in combination with sorafenib

INTERVENTIONS:
Drug: Treatment with ARQ 197 in combination with sorafenib — Patients will be treated with ARQ 197 and sorafenib at Dose Level 1 (ARQ 197 360 mg twice daily (bid) and sorafenib 200 mg bid). Patients with HCC will start treatment with ARQ 197 at 240 mg bid and sorafenib 200 mg bid. Enrollment of subsequent patient cohort will depend on the safety and tolerability of the combination treatment in the initial cohort.
  If < 33% patients treated at Dose Level 1 experience dose-limiting toxicity(ies) (DLT) by the end of first treatment cycle (4 weeks), then next cohort of 6 patients will be enrolled and treated at Dose Level 2 (ARQ 197 360 mg bid and sorafenib 400 mg bid). If ≥ 33% patients treated at Dose Level 1 experience DLT(s) by the end of first treatment cycle, the next cohort of 6 patients will be enrolled and treated at Dose Level 0 (ARQ 197 240 mg bid and sorafenib 200 mg bid).

SUMMARY:
This is an open-label, dose-escalation study of ARQ 197 administered orally in combination with sorafenib.

DETAILED DESCRIPTION:
The study is only enrolling patients in the expanded cohorts with hepatocellular carcinoma, renal cell carcinoma, melanoma, non-small cell lung cancer, and breast cancer.

Enrollment of an initial patient cohort of 3 or 6 patients will follow the traditional "3 + 3" dose escalation scheme. These patients will be treated with ARQ 197 and sorafenib at Dose Level 1 (ARQ 197 360 mg BID and sorafenib 200 mg BID). Enrollment of subsequent patient cohort(s) will depend on the safety and tolerability of the combination treatment in the initial cohort. If <33% patients treated at Dose Level 1 experience dose-limiting toxicity(ies) (DLT) by the end of first treatment cycle (4 weeks), then next cohort of 6 patients will be enrolled and treated at Dose Level 2 (ARQ 197 360 mg BID and sorafenib 400 mg BID). If ≥ 33% patients treated at Dose Level 1 experience DLT(s) by the end of first treatment cycle, the next cohort of 6 patients will be enrolled and treated at Dose Level 0 (ARQ 197 240 mg BID and sorafenib 200 mg BID).

Additional treatment cohorts may be enrolled to explore intermediate, higher or lower doses of ARQ 197, as indicated by the tolerability, safety profile, and pharmacokinetic (PK) profile.

Intra-patient dose-escalation from Dose Level 1 to Dose Level 2 may occur in patients enrolled in Dose Level 1 after they complete at least 1 cycle of treatment without DLT and other drug-related adverse event that, in the opinions of Investigator and Medical Monitor, is serious and medically significant.

Once a safe and recommended dose level is determined, an expanded cohort (Expansion Cohort 1) of up to 40 patients with either unresectable HCC or advanced renal cell carcinoma (RCC), for whom sorafenib is indicated, will be enrolled and treated at this dose level (expansion portion). Up to 20 patients with unresectable HCC and up to 20 patients with advanced RCC may be enrolled in this protocol (including patients in dose-escalation cohorts and expansion cohort).

An additional expansion cohort (Expansion Cohort 2) of up to 40 patients with breast cancer, non-small cell lung cancer or melanoma will be enrolled and treated at MTD/RP2D. Up to 10 patients may be enrolled for breast and non-small cell lung cancer and up to 20 patients with melanoma (at least 10 of whom must have NRAS mutation).

Under Amendment #3, newly enrolled subjects with HCC will be given ARQ 197 at 240 mg BID as starting dose. If a patient with HCC tolerates this starting dose for at least one cycle, the investigator may increase his/her dose to 360 mg BID.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent granted prior to initiation of any study-specific screening procedures
* 18 year of age or older
* Histologically or cytologically confirmed locally advanced, inoperable or metastatic solid tumors. In the two expansion cohorts, only patients with histologically or cytologically confirmed HCC, RCC, breast cancer, NSCLC and melanoma are eligible. An exception for this criterion is that patients with HCC may be enrolled without histological confirmation of disease so long as they meet the following criteria for diagnosis of HCC (and all other protocol eligibility criteria):

  1. Lesion > 2cm in diameter
  2. α-fetoprotein (AFP) > 200 ng/mL
  3. Radiological appearance of mass is suggestive of HCC
* Measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤1
* Adequate bone marrow, liver, and renal functions, defined as:
* Platelet count ≥ 100 × 10^9/L (≥ 60 × 10^9/L for HCC patients enrolled in the expanded cohort)
* Hemoglobin ≥ 10 g/dL
* Absolute neutrophil count (ANC) ≥1.5 × 10^9/L
* Total bilirubin ≤ 1.5 mg/dL or ≤ 3 mg/dL with HCC or metastatic liver disease
* Alanine transaminase (ALT) and aspartate transaminase (AST) ≤ 2.5 × upper limit of normal (ULN) or ≤ 5 × ULN with HCC or metastatic liver disease
* Serum creatinine ≤1.5 × ULN
* International normalized ratio (INR) 0.8 to 1.2 or 2 to 3 for patients receiving anticoagulant such as coumadin or heparin. Patients who are therapeutically anticoagulated are allowed to participate provided that no prior evidence of underlying abnormality exists in these parameters
* Women of childbearing potential must have a negative pregnancy test performed within seven days prior to the start of study drug
* Male and female subjects of child-bearing potential must agree to use double-barrier contraceptive measures, oral contraception, or avoidance of intercourse during the study and for 90 days after last investigational drug dose received

Exclusion Criteria:

* Previous anti-cancer chemotherapy, radiotherapy, immunotherapy or investigational agents within 4 weeks prior to the first day of study defined treatment with the following exceptions: 1) a prostate cancer patient on androgen deprivation with gonadotropin-releasing hormone (GnRH) agonists can be enrolled while he remains on the immunotherapy; 2) a patient received palliative radiotherapy previous can be enrolled if the therapy was completed 1 week (7 days) prior to the first day of study defined treatment and the patient has recovered from any radiotherapy-related adverse event(s); and 3) patients are currently on sorafenib can be enrolled
* History of cardiac disease: congestive heart failure defined as Class II to IV per New York Heart Association (NYHA) classification; active coronary artery disease (CAD); previously diagnosed clinically significant bradycardia, other uncontrolled cardiac arrhythmia defined as ≥ Grade 2 according to National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) (version 3.0), or uncontrolled hypertension; myocardial infarction occurred within 6 months prior to study entry (myocardial infarction occurred > 6 months prior to study entry is permitted)
* Active clinically serious infections defined as ≥ Grade 2 according to NCI CTCAE, version 3.0
* Substance abuse, medical, psychological or social conditions that may, in the opinion of the Investigator, interfere with the patient's participation in the study or evaluation of the study results
* Any condition that is unstable or which could jeopardize the safety of the patient and his/her protocol compliance
* Known human immunodeficiency virus (HIV) infection
* Pregnancy or breast-feeding
* Inability to swallow oral medications
* Significant gastrointestinal disorder, in the opinion of the Investigator, could interfere with the absorption of ARQ 197 and/or sorafenib (e.g. significant, uncontrolled inflammatory bowel disease or extensive small bowel resection).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2009-09; Primary Completion 2012-09 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
To identify maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D) of ARQ 197 when administered in combination with sorafenib. | 6 to 9 months. Patients will remain on study until progression of disease, unacceptable toxicity, or other discontinuation criterion is met.

SECONDARY OUTCOMES:
To determine the pharmacokinetic profiles of ARQ 197 and sorafenib. | Patients will remain on study until progression of disease, unacceptable toxicity, or other discontinuation criterion is met.
To assess the preliminary anti-tumor activity of ARQ 197 when administered in combination with sorafenib. | Patients will remain on study until progression of disease, unacceptable toxicity, or other discontinuation criterion is met.
To evaluate dynamic changes of hepatocyte growth factor (HGF), vascular endothelial growth factor (VEGF), and soluble c-Met in patients' peripheral blood that are associated with treatment of ARQ 197 plus sorafenib. | Patients will remain on study until progression of disease, unacceptable toxicity, or other discontinuation criterion is met.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (3):
  - Boston, Massachusetts
  - Roswell Park Cancer Institute, Buffalo, New York
  - Nashville, Tennessee
- Rozzano, Italy